CLINICAL TRIAL: NCT07141095
Title: A Prospective Single-Arm Observational Study of Maribavir for the Treatment of Post Hematopoietic Stem Cell Transplantation Cytomegalovirus Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2025003
Record Dates: First submitted 2025-07-30; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Infections, Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — maribavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CMV Infection: Participants will receive maribavirv tablets, 400 mg, orally twice a day(bid) for up to 8 weeks treatment period.
  Interventions: Drug: maribavir

INTERVENTIONS:
Drug: maribavir — Maribavir tablets are administered orally at a dose of 0.4 g per administration (2 tablets of 0.2 g each), twice daily. The recommended duration of treatment is 8 weeks; however, the specific treatment duration should be individualized based on the clinical characteristics of each patient.

SUMMARY:
The main aim of this study is to check the effectiveness and safety of maribavir for the treatment of CMV infection after HSCT in Chinese patients in real-world settings.

The participants will be treated with maribavir for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic Stem Cell Transplant Recipients

  1. Adult patients with an expected survival of ≥4 weeks.
  2. Confirmed CMV infection, including CMV viremia and CMV disease.
  3. Fully understand the content of the trial, voluntarily participate and complete the trial, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Participants who meet any of the following criteria are not eligible for this study:

  1. Patients currently participating in other CMV-related clinical studies, such as those receiving anti-CMV drug treatment or involved in CMV vaccine clinical studies.
  2. At screening, liver function tests show: AST > 5×ULN, or ALT > 5×ULN, or total bilirubin ≥ 3.0×ULN.
  3. Patients with psychiatric disorders or severe psychological conditions that may affect the ability to provide informed consent or participate in follow-up consultations.
  4. Participants deemed unsuitable for inclusion by the investigator.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed CMV infection, including CMV viremia and CMV disease after Hematopoietic Stem Cell Transplant.
Sampling Method: Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
CMV viremia clearance rate | At Week 4
  The proportion of patients who had confirmed clearance of CMV viremia in plasma (defined as two consecutive CMV-DNA tests below the preemptive treatment threshold after treatment) after 4 weeks of treatment.
CMV disease remission rate | At Week 4
  The proportion of patients who achieved remission of CMV disease after 4 weeks of treatment.

SECONDARY OUTCOMES:
Number of participants with AEs | From first dose of study drug up to week 8
  An AE was defined as any event emerging or manifesting at or after the initiation of treatment with a medicinal product or any existing event that worsened in either intensity or frequency following exposure to the medicinal product.
CMV DNA undetected time | From first dose of study drug up to week 8
  The time when CMV DNA was first detected under the limit of detection in plasma.
CMV viremia clearance at the end of 8 weeks of treatment | At Week 8
  The proportion of patients with confirmed clearance of CMV viremia in plasma at the end of 8 weeks of treatment.
Number of participants with all-cause mortality | From first dose of study drug up to week 8
  All-cause mortality means death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China